CLINICAL TRIAL: NCT04265443
Title: Prognostic Perspective of Invasive Hyperemic and Non-Hyperemic Physiologic Indices Measured After Percutaneous Coronary Intervention (PERSPECTIVE-PCI)
Brief Title: Prognostic Perspective of Invasive Hyperemic and Non-Hyperemic Physiologic Indices Measured After Percutaneous Coronary Intervention
Acronym: PERSPECTIVEPCI
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Inje University Ilsan Paik Hospital (Other); Ulsan University Hospital (Other); Sejong General Hospital (Other); Chosun University Hospital (Other)
Responsible Party: Principal Investigator, Joo Myung Lee, Assistant Professor, Samsung Medical Center
Other Study IDs: POSTPCI_NHPRs20200206
Record Dates: First submitted 2020-02-06; First posted 2020-02-11 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Ischemic Heart Disease
Keywords: fractional flow reserve; non-hyperemic pressure ratio; percutaneous coronary intervention; prognosis; myocardial ischemia
MeSH Terms: conditions — Myocardial Ischemia | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post PCI state: The study population of this study underwent percutaneous coronary intervention(PCI) with 2nd generation drug-eluting stent (DES) and measured invasive physiologic indices after PCI
  Interventions: Device: Percutaneous coronary intervention

INTERVENTIONS:
Device: Percutaneous coronary intervention — PCI was performed using 2nd generation DES

SUMMARY:
Coronary physiologic assessments by the pressure-derived fractional flow reserve (FFR) have become standard methods for identifying hemodynamic deprivation in coronary arterial stenosis for evidence-based percutaneous coronary intervention (PCI). Invasive physiologic indices-guidance enables on-site real time assessment for functional significance of epicardial coronary stenosis and the use of those indices has shown to be effective to guide treatment decision. Several studies further support the role of post-PCI FFR measurement as a functional marker of residual disease after PCI and prognostic indicator of patients. Although optimal cut-off values of post-PCI FFR varied across studies, an inverse relationship between post-PCI FFR and the risk of future clinical events have been reported consistently.

Recently, non-hyperemic pressure ratios (NHPRs) have been introduced in clinical practice. Although there are several different NHPRs, previous studies consistently indicated that those NHPRs shares similar diagnostic performance and prognostic implications. Nevertheless, few reports were available for clinical relevance of NHPRs in evaluation of post-PCI status.

In this context, we will evaluate the physiologic characteristics and prognostic implication of post-PCI NHPRs and compare with those of post-PCI FFR in patients who underwent angiographically successful PCI with 2nd generation drug-eluting stent implantation (DES).

DETAILED DESCRIPTION:
Patients who diagnosed significant coronary artery disease and treated by 2nd generation DES with post-PCI physiologic evaluation would be enrolled.

Invasive physiologic assessment including recording of resting pressure trecing would be required at the baseline and at the end of index PCI procedure. PCI procedure would be performed upon local routine. Any available 2nd generation DES could be used. Web-based electronic-case record form (CRF) system will be used for collecting data. All data will be handled and analyzed by blind fashion at independent core lab. 2-year clinical outcome after index procedure will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* any patient meets eligible criteria who underwent PCI with DES followed by invasive physiologic assessment at the index procedure
* available both post-PCI resting pressure tracing and FFR

Exclusion Criteria:

* culprit vessel of acute coronary syndrome
* failed achieving TIMI 3 flow at the end of PCI
* left ventricular ejection fraction <30%
* graft vessel
* collateral feeder
* in-stent restenosis
* primary myocardial or valvular heart disease
* in patient whose life expectancy less than 2 years
* visible thrombus of target vessel segment
* unmeasured post-PCI resting pressure tracings

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who diagnosed obstructive coronary artery disease and treated by DES with invasive physiologic evaluation at the index procedure
Sampling Method: Non-Probability Sample
Enrollment: 588 (Actual)
Dates: Start 2013-05-13 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Target Vessel Failure | 2 years after index procedure
  a composite of cardiac death, clinically-driven target vessel-related myocardial infarction, and clinically-driven target vessel revascularization. The target vessel will be defined as the treated vessel with 2nd generation DES which was assessed by post stent fractional flow reserve.

SECONDARY OUTCOMES:
independent predictors for target-vessel failure | 2 years after index procedure
  independent predictors for target-vessel failure by univariate and multivariate analysis will be performed.
delta FFR per unit time | At the time of index procedure
  delta FFR per unit time in pre-PCI pullback recording
Relative percent increase of physiologic indices | At the time of index procedure
  Percent increase of FFR or non-hyperemic pressure ratios

CONTACTS AND LOCATIONS:
Overall Officials: Joo Myung Lee, MD, MPH, PhD, Principal Investigator — Samsung Medical Center
Locations (5):
- South Korea (5):
  - Sejong General Hospital, Bucheon-si
  - Inje University Ilsan Paik Hospital, Goyang-si
  - Chosun University Hospital, Gwangju
  - Samsung Medical Center, Seoul
  - Ulsan Medical Center, Ulsan

IPD SHARING:
Plan to Share IPD: Undecided
De-identified patient data will be shared upon reasonable request after discussion in executive committee.

REFERENCES:
- [Derived] Lee JM, Joh HS, Choi KH, Hong D, Park TK, Yang JH, Song YB, Choi JH, Choi SH, Jeong JO, Lee JY, Choi YJ, Chae JK, Hur SH, Bae JW, Oh JH, Chun KJ, Kim HJ, Cho BR, Shin D, Lee SH, Hwang D, Lee HJ, Jang HJ, Kim HK, Ha SJ, Shin ES, Doh JH, Hahn JY, Gwon HC; SMART-REWARD Investigators. Safety and Efficacy of Everolimus-Eluting Bioresorbable Vascular Scaffold Versus Second-Generation Drug-Eluting Stents in Real-World Practice. J Korean Med Sci. 2023 Feb 6;38(5):e34. doi: 10.3346/jkms.2023.38.e34. PMID 36747363
- [Derived] Shin D, Lee SH, Lee JM, Choi KH, Hwang D, Lee HJ, Jang HJ, Kim HK, Kwak JJ, Ha SJ, Song YB, Shin ES, Doh JH. Prognostic Implications of Post-Intervention Resting Pd/Pa and Fractional Flow Reserve in Patients With Stent Implantation. JACC Cardiovasc Interv. 2020 Aug 24;13(16):1920-1933. doi: 10.1016/j.jcin.2020.05.042. PMID 32819481